CLINICAL TRIAL: NCT06035887
Title: A Feasibility Study Using Novel, Portable Electroretinography Devices to Detect Hydroxychloroquine Retinopathy
Brief Title: Novel ERG for Detection of Hydroxychloroquine Retinopathy
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: LUPUS UK (Unknown); King's College Hospital Charity (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS 317611
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Hydroxychloroquine Retinopathy
Keywords: Electroretinography; Diagnostic Evaluation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Normative Controls: Age- and sex- matched normal controls
  Interventions: Diagnostic Test: Hand-Held Full-Field Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Trolley-Mounted Multifocal Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Spectral-Domain Optical Coherence Tomography (Standard of Care test); Diagnostic Test: Macular Autofluorescence (Standard of Care test)
- On Hydroxychloroquine, NO retinopathy: Participants over 18 years on hydroxychloroquine without hydroxychloroquine-related retinopathy
  Interventions: Diagnostic Test: Hand-Held Full-Field Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Trolley-Mounted Multifocal Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Spectral-Domain Optical Coherence Tomography (Standard of Care test); Diagnostic Test: Macular Autofluorescence (Standard of Care test)
- On Hydroxychloroquine, POSSIBLE retinopathy: Participants over 18 years on hydroxychloroquine with possible (indeterminate) hydroxychloroquine-related retinopathy
  Interventions: Diagnostic Test: Hand-Held Full-Field Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Trolley-Mounted Multifocal Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Spectral-Domain Optical Coherence Tomography (Standard of Care test); Diagnostic Test: Macular Autofluorescence (Standard of Care test)
- On Hydroxychloroquine, DEFINITE retinopathy: Participants over 18 years on hydroxychloroquine with definite hydroxychloroquine-related retinopathy
  Interventions: Diagnostic Test: Hand-Held Full-Field Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Trolley-Mounted Multifocal Skin-Electrode Electroretinography (Device to be evaluated); Diagnostic Test: Spectral-Domain Optical Coherence Tomography (Standard of Care test); Diagnostic Test: Macular Autofluorescence (Standard of Care test)

INTERVENTIONS:
Diagnostic Test: Hand-Held Full-Field Skin-Electrode Electroretinography (Device to be evaluated) — RETEval Complete hand-held electroretinogram
Diagnostic Test: Trolley-Mounted Multifocal Skin-Electrode Electroretinography (Device to be evaluated) — UTAS multifocal electroretinogram
Diagnostic Test: Spectral-Domain Optical Coherence Tomography (Standard of Care test) — Heidelberg Engineering Spectralis Spectral-Domain Optical Coherence Tomography (macular structural scan)
Diagnostic Test: Macular Autofluorescence (Standard of Care test) — Heidelberg Engineering Spectralis Autofluorescence imaging (macular structural image)

SUMMARY:
The purpose of the study is to investigate novel electroretinography (ERG) devices in the detection of hydroxychloroquine retinopathy. Two devices (the RETEval full-field and flicker ERG and UTAS multifocal ERG) will be evaluated in this study, comparing device outputs to standard of care screening tests, in groups of participants characterised by presence or absence of hydroxychloroquine-related retinopathy.

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ) is a widely used drug used to treat disorders of inflammation in the body with up to 320,000 people estimated to be on this drug in the UK alone. Retinopathy due to HCQ is a significant problem, necessitating yearly screening which can only realistically take place in hospital eye units where funding and capacity constraints limit the provision of services.

Electroretinography is a non-invasive method of testing for eye retinal problems, which works by flashing light (in certain patterns and brightness) into eyes and measuring the electrical response through fine wires placed on the eye surface or behind the eyelid, and is considered by many authors to be a gold-standard test to detect HCQ retinopathy. Their use has been limited due to the high expertise required to undertake and interpret tests, limited availability of testing, and high test burden, however newer electroretinography devices have been developed by a company called LKC Technologies, which are faster to perform, use leads placed on the skin (rather than the eye surface) which are more comfortable, easier to use by healthcare technicians, and can be done without the need for dilating eyedrops. The two devices being tested in this study are:

* The RETEval = a handheld electroretinography testing device
* The UTAS multifocal ERG = a trolley-mounted electroretinography testing device

These innovations may make testing far easier to develop in both hospital eye service, and potentially even general settings such as outpatient clinics, general practices, and optometrists. This study aims to evaluate the performance of devices to detect and classify participants in 4 main groups:

* Normative control participants (n=35)
* Patients taking HCQ but without retinopathy (n=35)
* Patients taking HCQ with indeterminate features of retinopathy (also known as POSSIBLE retinopathy) (n=35)
* Patients taking HCQ with definite retinopathy

Device outputs will be analysed and compared with masked graded screening results (incorporating spectral-domain macular optical coherence tomography and autofluorescence as standard, taken on the same visit) to generate device- and device-output-specific sensitivities and specificities. If a signal is found, the feasibility outcomes from this study will inform the study methodology and timelines for a larger trial if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. HCQ groups:

   a. HCQ use >5 years for patients without any high-risk factors, or >1 year in patients with one or more high-risk factors for HCQ retinopathy, namely: i. Dose >5mg/kg per day actual body weight (ABW) ii. Estimated glomerular filtration rate (eGFR) of <60mls/min/1.73m2 iii. Concomitant tamoxifen use
3. Control group:

   1. No prior HCQ exposure

Exclusion Criteria:

1. Cataract grade ≥3 of any subtype
2. Recent cataract surgery within 4 weeks of recruitment
3. Significant media opacity or corneal disease including, but not limited to, corneal oedema, corneal scarring, keratoconus, previous corneal transplants, severe keratoconjunctivitis sicca (requiring the use of topical serum, immunosuppressive or analogous therapy, or procedural treatment).
4. Significant macular co-pathology including, but not limited to, macular degeneration, macular scarring, cystic macular oedema (for any reason), staphyloma.
5. Inherited retinal and/or macular dystrophies including colour vision deficiencies
6. Active or previous posterior uveitis or pan-uveitis
7. Aphakia
8. High refractive error >6.00 dioptres
9. Amblyopia
10. Diabetes
11. Retinal angiopathies including, but no limited to, retinal vein occlusion, retinal artery occlusion, ocular ischaemic syndrome, HIV retinopathy, Sickle cell disease, radiation retinopathy
12. Visually significant surgical retinal disease including epiretinal membrane, macular hole, retinal detachment, retinal tear
13. Previous retinal laser or intravitreal treatment
14. Moderate or worse glaucoma
15. Optic atrophy
16. Photosensitive epilepsy
17. Ungradable HCQ retinopathy screening images
18. Periocular infection or rash (recruitment can be deferred until acute pathology has resolved)
19. Unable or unwilling to undertake study activities
20. Any active use or history of the following medications:

Amiodarone Canthaxanthin Deferoxamine Digoxin Ethambutol Interferon-alpha Melatonin Nefazodone Sildenafil Vigabatrin Chloroquine Quinine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Age- and sex-matched control group (n=35) On hydroxychloroquine without retinopathy (n=35) On hydroxychloroquine with possible retinopathy (n=35) On hydroxychloroquine with definite retinopathy (n=35)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of both devices to discriminate between NO, POSSIBLE and DEFINITE hydroxychloroquine retinopathy compared to standard screening tests | All tests required to determine sensitivity and specificity of both devices compared to standard retinal imaging will be completed in a single visit. Safety will be evaluated up to 1 week post-visit.
  Primary Outcome

SECONDARY OUTCOMES:
To compare the sensitivity and specificity of undilated versus dilated testing with the multifocal ERG device, for all categories of hydroxychloroquine retinopathy | All tests required to determine this outcome will be completed at a single visit. Safety will be evaluated up to 1 week post-visit.
  Secondary Outcome
To determine the patient acceptability of both devices evaluated using standardised, study-specific questionnaires | All tests required to determine this outcome will be completed at a single visit. Safety will be evaluated up to 1 week post-visit.
  Feasibility Outcome
To determine the proportion and recruitment rate of patients in each category of hydroxychloroquine retinopathy who consent to join this study. | All tests required to determine this outcome will be completed at a single visit. Safety will be evaluated up to 1 week post-visit.
  Feasibility Outcome

OTHER OUTCOMES:
To determine which ERG waveform features (such as implicit time or amplitude) from both devices best discriminate participants with NO hydroxychloroquine retinopathy from those with POSSIBLE and DEFINITE hydroxychloroquine retinopathy | All tests required to determine this outcome will be completed at a single visit. Safety will be evaluated up to 1 week post-visit.
  Exploratory Outcome
To determine if both device waveforms correlate with standard mfERG waveforms in patients receiving hydroxychloroquine | All tests required to determine this outcome will be completed at a single visit. Novel device ERG waveforms will be compared with standard mfERG where undertaken in the preceding 12 months. Safety will be evaluated up to 1 week post-visit.
  Exploratory Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Professor Timothy L Jackson, Study Chair — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee CN, Wafa HA, Murphy G, Galloway J, Mahroo OA, Jackson TL. Novel electroretinography devices to detect hydroxychloroquine retinopathy: study protocol for a diagnostic accuracy and feasibility study. BMJ Open Ophthalmol. 2024 Dec 24;9(1):e001898. doi: 10.1136/bmjophth-2024-001898. PMID 39719323